CLINICAL TRIAL: NCT06348979
Title: Clinical Performance of Fiber Reinforced FRC Base and Bonded CAD/CAM Resin Composite Endocrowns Versus Conventional Lithium Disilicate Endocrowns in Posterior Teeth (1y Randomized Clinical Trial)
Brief Title: Clinical Performance of Fiber Reinforced FRC Base and Bonded CAD/CAM Resin Composite Endocrowns
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Sherifa Ahmed Abdelaziz Kandil, Lecturer, Conservative dentistry department, Faculty of Dentistry, Cairo University., Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CEBD 5/2021
Record Dates: First submitted 2023-12-07; First posted 2024-04-05 (Actual); Last update posted 2024-04-05 (Actual); Status verified 2024-03

CONDITIONS: Dental Caries
Keywords: restoration fracture; CAD/CAM resin composite endocrowns; lithium disilicate endocrowns
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hybrid Nano-ceramic (Grandio) CAD/CAM Endocrowns (Experimental): Adding of short fiber reinforced flowable resin composite material (everX Flow, GC Europe) as a supporting base under CAD/CAM resin composite endocrowns
  Interventions: Procedure: Fiber flowable (SFRC) support below hybrid nanoceramic endocrowns
- Lithium Disilicate (e.max) Endocrowns (Active Comparator): Lithium Disilicate (e.max) Endocrowns
  Interventions: Procedure: all ceramic Endocrowns (emax)

INTERVENTIONS:
Procedure: Fiber flowable (SFRC) support below hybrid nanoceramic endocrowns — restoration of endodontically treated teeth by endocrowns
  Other Names: Grandio CAD/CAM block
  Arms: Hybrid Nano-ceramic (Grandio) CAD/CAM Endocrowns
Procedure: all ceramic Endocrowns (emax) — restoration of endodontically treated teeth by endocrowns
  Arms: Lithium Disilicate (e.max) Endocrowns

SUMMARY:
This research proposal is introduced to clinically test short fiber reinforced flowable resin composite material (everX Flow, GC Europe) as a supporting base under CAD/CAM resin composite endocrowns due to gap of knowledge present in this area.

ELIGIBILITY:
Inclusion Criteria:

* Endodontically treated molar teeth indicated for endocrown.
* Presence of favorable occlusion and teeth are in normal alignment with the adjacent teeth, -medically free

Exclusion Criteria:

* ▪ Endodontically treated molar teeth indicated for post and core or only crown coverage.

  * Severe periodontal problems

Ages: 18 Years to 38 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 110 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2024-01-30 (Actual)

PRIMARY OUTCOMES:
clinical Fracture | change from baseline and months: 3, 6, 12
  modified usphs criteria (alpha, bravo, charlie) with measuring unit: scoring system (ordinal)

SECONDARY OUTCOMES:
clinical performance marginal adaptation | change from baseline and months: 3, 6, 12
  modified usphs criteria (alpha, bravo, charlie) with measuring unit:scoring system (ordinal)

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No